CLINICAL TRIAL: NCT03396549
Title: Effect of tDCS Montage on Measures of Appetite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Mary Boggiano, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB-300000049
Record Dates: First submitted 2017-12-28; First posted 2018-01-11 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Eating Behavior
Keywords: tDCS; food craving; tDCS sham procedure; montage; food intake
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Cross-over blind. All get sham and real tDCS.
Who Masked: Participant, Outcomes Assessor
Masking Description: Only the assistant delivering tDCS will not be blind to conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real tDCS (Experimental): 20 min of 2 mA tDCS over the right and left dorsolateral prefrontal cortex
  Interventions: Device: real tDCS
- new sham tDCS (Sham Comparator): 20 min 2 mA tDCS over the left and right sensorimotor cortex
  Interventions: Device: new sham tDCS

INTERVENTIONS:
Device: new sham tDCS — 1 ch TCT transcranial stimulator
  Arms: new sham tDCS
Device: real tDCS — 1 ch TCT transcranial stimulator
  Arms: real tDCS

SUMMARY:
The aim is to validate a new sham (control) method for use in transcranial direct current stimulation (tDCS) that is less discernible to participants from the real condition. Participants are often able to tell real from sham conditions. Correctly guessing real from sham undermines the integrity of evaluations of the value of tDCS as a treatment tool as responses may be in part or entirely the result of treatment expectation effects. The study will test a new sham method to reduce food craving and eating and test how much participants are able to discern it from the real or 'target' condition.

DETAILED DESCRIPTION:
On Visit One:

N=30 college students will be given a unique assigned ID# to use on all electronic surveys. A Face Sheet will also record how hungry they feel at the time and will be rescheduled if overly hungry or full. Participants will then be measured for a BMI.

Participants will then complete an electronic survey that includes demographic questions including age, sex, ethnicity, handedness, and if they are vegan or vegetarian (to dismiss craving responses on animal-based foods on the food craving task). This is followed by an electronic battery of psychological questionnaires to assess eating motives, binge-eating, dietary restraint, impulsiveness, and suggestibility. Participants will then complete the Food Craving Task. They will do this immediately before and immediately after the tDCS session. Before the tDCS session participants will be shown a series of 24 colored images of appealing foods on the computer monitor and will be asked to rate how much they "like" the food and to measure craving: "how much they would like to eat the food right now if it were available" using a rating scale. After the tDCS session participants will be shown the same 24 photos and asked to rate them only for craving, not liking, as tDCS is not expected to change liking of foods. Liking ratings are taken so that only liked foods (rated a 2, 3, or 4 on the scale) are analyzed for their craving (wanting) scores. This avoids erroneous interpretation of decreased craving for the foods as being due to tDCS when the real reason is that they were not liked to begin with. Participants will then be escorted to the tDCS and eating room where they will then be seated in a comfortable chair facing a table a few yards away with three plates of food for the eating task. The researcher administering tDCS will instruct them to relax while she/he takes head measurements with a measuring tape. The measurements are taken according to the EEG 10-20 system to locate F3 and F4 which correspond to the left and right dorsolateral prefrontal cortex (DLPFC), or C3 and C4 which correspond to the left and right somatosensory/sensorimotor cortex (SSSM), depending on which montage they are receiving on the first visit. For the DLPFC, the anode will be placed over the right and cathode over the left DLPFC. For the SSSM, the anode will be placed over the left and cathode over the right SSSM. Two researchers will be present to facilitate the head measurements and confirm the accuracy of electrode placement. The locations are marked with a Sharpie marker on the scalp. The two 35 mm2 electrodes are covered in sponge sleeves with saline solution. These are placed over the marked locations and held by an adjustable head band. The researcher will turn on the device which will ramp up to 2 milliamps (mA) current in 30 seconds, hold at 2mA for 19 minutes them ramp down in the last 30 seconds for a total stimulation time of 20 minutes. During the session participants will be handed the Physical Sensations Scale (PSS) to rate sensation types and intensity for the first 5, 10, 15, and last minute of the session. The PSS is a modified version from Clark et al., 2012, and has been used successfully in Boggiano's previous tDCS studies. The modified PSS provides ratings that are more sensitive and individualized and will be submitted for publication consideration. They will know from reading the Consent Form and the PSS the possible sensations they may experience. The scale will be completed more times than the usual 1-2 times per session because it will be used to evaluate differences in sensations between the two tDCS montages. Low to no differences will indicate a good sham for the DLPFC montage. Immediately following the tDCS session, they will go back to the computer room to complete the post-tDCS part of the Food Craving Task as described above. After this, participants will be escorted back to the tDCS/eating room and will be given 15 minutes to consume the foods displayed on the table. The participants will then be escorted back to the computer room for a last Visit 1 Post-Eating Questionnaire. This is intended to obtain more information about any perceived changes in appetite or other functions following tDCS and compare them across the two montages.

On Visit Two:

As in Visit One, participants will then complete another pre-tDCS Food Craving Task with only the wanting questions as their liking of the foods on the photos is not expected to change. They will then receive the alternate tDCS montage as described for Visit One and complete the PSS four times during the session, followed by the post-tDCS Food Craving Task and another In-Lab Eating Task and "Visit 2 Post-Eating Questionnaire". This one will be exactly like the Visit 1 Post-Eating Questionnaire except that it will also ask participants to rank the 3 foods from most to least preferred in order to obtain the added measures of preferred-food eaten (mean of the #1-ranked food kcals) and less-preferred food eaten (mean of the average kcals between the #2- and #3-ranked foods). The researcher will then conduct a person-to-person omnibus interview with the Real vs. Sham Interview (RSI). This is designed to help validate the new sham method using the participants' perceptions of both sessions. The participants are then debriefed and compensated the participant.

ELIGIBILITY:
Inclusion Criteria:

* UAB student
* Age 18-55

Exclusion Criteria:

* Implanted cranial metal plates or medical devices
* History of brain surgery
* Loss of consciousness > 5 minutes
* Post-trauma amnesia lasting more than 30 minutes
* Diagnosis of schizophrenia, bipolar disorder, bulimia nervosa, anorexia nervosa, depression with suicidal intent or ideation
* Enrollment in a commercial weight-loss program
* Pregnancy or breastfeeding
* Uncontrolled diabetes or hypertension
* Current illicit drug use
* Intent to stop or begin use of a prescription drug or drugs that influence appetite
* Allergy to ingredients in the food that will be used in the eating test (e.g., wheat, gluten, soy, chocolate).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2018-03-14 (Actual); Study Completion 2018-03-14 (Actual)

PRIMARY OUTCOMES:
Eating Behaviors | 20 minutes
  Amount of food eaten in kcals and food craving in ratings for degree of wanting a particular food displayed on computer screen.

SECONDARY OUTCOMES:
Detection of target from sham tDCS session. | 20 minutes
  Difference between physical sensation ratings felt during the session and likert-like response ratings to an interview.

CONTACTS AND LOCATIONS:
Overall Officials: Mary M Boggiano, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham (UAB), Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No